CLINICAL TRIAL: NCT00645099
Title: A Prospective Randomized Open-label 6-Month Head-To-Head Trial to Compare Metabolic Effects of Paliperidone ER and Olanzapine in Subjects With Schizophrenia
Brief Title: A 6 Month Study to Compare the Metabolic Effects of Paliperidone ER and Olanzapine in Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR013189; R076477SCH3020
Record Dates: First submitted 2008-03-24; First posted 2008-03-27 (Estimated); Results first posted 2010-07-29 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-04

CONDITIONS: Schizophrenia
Keywords: Paliperidone ER; Olanzapine; Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Olanzapine; Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 001 (Experimental): paliperidone ER 6-mg or 9-mg tablet once daily flexible dosing for 6 months
  Interventions: Drug: paliperidone ER
- 002 (Active Comparator): olanzapine 10-15 mg (using 5-mg or 10-mg tablets) once daily flexible dosing for 6 months
  Interventions: Drug: olanzapine

INTERVENTIONS:
Drug: olanzapine — 10-15 mg (using 5-mg or 10-mg tablets) once daily flexible dosing for 6 months
  Arms: 002
Drug: paliperidone ER — 6-mg or 9-mg tablet once daily flexible dosing for 6 months
  Arms: 001

SUMMARY:
The purpose of this 6 month study is to compare the metabolic effects of paliperidone ER and olanzapine in patients with schizophrenia, using the ratio of the concentration of lipids (triglycerides (TG)) in the blood to the concentration of good cholesterol (high density lipoproteins (HDL)) in the blood as the primary parameter. Approximately 456 adult patients will participate in this study.

DETAILED DESCRIPTION:
This is a prospective randomized (study medication is assigned by change) open-label, parallel-group, multicenter, 6 month study to compare the metabolic effects of paliperidone ER and olanzapine in patients with schizophrenia using the ratio of the concentration of lipids (triglycerides) in the blood to the concentration of good cholesterol (high density lipoproteins (HDL)) as the primary parameter. Secondary objectives include evaluation of additional parameters related to the total of the actions of the body to keep it alive (metabolic endpoints) and demonstration of non-inferiority of paliperidone ER versus olanzapine in efficacy as measured by Positive and Negative Syndrome Scale (PANSS). Patients previously treated with any oral antipsychotic, except those treated with paliperidone ER, olanzapine or clozapine during the last 6 months, can be enrolled and will be treated with paliperidone ER (6 to 9 mg/day) or olanzapine (10 to 15 mg/day). Patients will be divided into groups according to the metabolic effects of their previous antipsychotic medication (medication that does not increase body weight vs. medication that increases body weight). Throughout the study flexible dosing is allowed based on the investigator discretion. A study treatment period of 6 months is planned for all patients. Medication to treat symptoms like confusion, blurred vision, constipation, dry mouth, light-headedness, difficulty starting and continuing to urinate, and loss of bladder control may continue up to four weeks and should then be tapered off at the discretion of the investigator. Approximately 456 adult patients (228 in each treatment group) will participate in this study. Efficacy will be assessed with the following measures: PANSS (total score and subscale scores), Clinical Global Impression - Severity (CGI-S), Self-rated health status Survey SF-36, and Sleep and daytime drowsiness evaluation scale. The parameters related to the total of the actions of the body to keep it alive (metabolic endpoints) will be assessed with the following: ratio of blood lipids to blood good cholesterol concentrations (TG:HDL ratio) (for this primary evaluation, plasma fasting lipids and good cholesterol concentrations will be measured), fasting plasma insulin and fasting plasma glucose, plasma glucose and insulin concentrations before and after a 75 gram oral glucose tolerance test (OGTT) to asses insulin sensitivity and changes in insulin secretion, fasting good cholesterol, lipids, and glucose levels for the determination of new onset or presence of metabolic syndrome during treatment according to criteria of the Third Report of the National Cholesterol Education Program Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (NCEP/ATPIII criteria), weight, Body-Mass-Index and waist circumference for the determination of new onset or presence of a medical condition associated with abdominal obesity, abnormalities in glucose, lipid and cholesterol metabolism, and elevated blood pressure that increases the risk of cardiovascular disease and type 2 diabetes (metabolic syndrome) during treatment according to NCEP/ATP III criteria. All patients who receive trial medication (paliperidone ER or olanzapine) at least once will be included in the analysis of the demographic and baseline characteristic data. 2 dosage levels of paliperidone ER (6 or 9mg per day) and 2 of olanzapine (10 and 15mg per day) are available to the patients. Throughout the study flexible dosing is allowed based on the investigator's discretion. Study medication is to be taken in the morning orally, with water. A study treatment period of 6 months is planned for all patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient meets the DSM-IV criteria for schizophrenia
* Patient has a PANSS total score at screening of 60 to 100, inclusive
* Patient must, in the opinion of the investigator, benefit from treatment with paliperidone ER or olanzapine
* Patients on lipid-lowering therapy must be on a stable dose for at least 4 weeks for statins, niacin, ezetimibe and resins or for at least 12 weeks for fibrates
* Female patients must be postmenopausal (for at least 1 year), surgically sterile, abstinent, or, if sexually active, be practicing and effective method of birth control (e.g. prescription oral contraceptives, contraceptive injections, intrauterine device, double-barrier method, contraceptive patch, male partner sterilization) before entry and throughout the study
* Women of child-bearing potential must have a negative urine pregnancy test at screening
* Patient is healthy on the basis of a physical examination and vital signs at screening

Exclusion Criteria:

* Patient has previously been treated with paliperidone ER, olanzapine, or clozapine within the past 6 months or has never been treated with an antipsychotic before
* Treatment with a depot antipsychotic within the past 3 months
* Treatment with a mood stabilizer or a recently initiated antidepressant (<= 3 months)
* Patient has abnormal fasting plasma glucose (> 126 mg/dL) or fasting triglycerides (TG) levels (> 400 mg/dL) at screening
* Relevant history of any significant and/or unstable cardiovascular, respiratory, neurologic (including seizures or significant cerebrovascular), renal, hepatic, endocrine, or immunologic diseases, including recent or present clinically relevant laboratory abnormalities (as deemed by the investigator)
* History or current symptoms of tardive dyskinesia
* History of neuroleptic malignant syndrome
* Pregnant or breast-feeding female

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Actual)
Dates: Start 2007-10; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (46):
- Argentina (3):
  - Buenos Aires
  - Córdoba
  - Mendoza
- Egypt (3):
  - Alexandria
  - Cairo
  - El Banfaig 2 District
- Estonia (3):
  - Pärnu
  - Tallinn
  - Tartu
- France (5):
  - Allonnes
  - Bron
  - Dijon
  - Limoges
  - Montberon
- Athens, Greece
- Amman, Jordan
- Latvia (5):
  - Jelgava
  - Liepāja
  - Riga
  - Sigulda
  - Strenči
- Beirut, Lebanon
- Lithuania (2):
  - Kaunas
  - Vilnius
- Romania (5):
  - Cluj-Napoca
  - Craiova
  - Oradea
  - Sibiu
  - Tg Mures
- Slovakia (3):
  - Bratislava
  - Michalovce
  - Rimavská Sobota
- South Africa (2):
  - Cape Town
  - Johannesburg
- Spain (8):
  - A Coruña
  - Alicante
  - Barcelona
  - Elche
  - Madrid
  - Santander
  - Vic
  - Zamora
- Turkey (Türkiye) (4):
  - Ankara
  - Bursa
  - Istanbul
  - Manisa

REFERENCES:
- See also: A Prospective Randomized Open-label 6-Month Head-To-Head Trial to Compare Metabolic Effects of Paliperidone ER and Olanzapine in Subjects With Schizophrenia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=50&filename=CR013189_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three subjects of the 462 enrolled did not receive study medication and were excluded from analysis: 2 subjects were randomized by mistake by the investigator and 1 subject withdrew consent before first intake of study medication. The ITT population consisted of 459 subjects who took at least one dose of study medication.
Groups:
- Paliperidone Extended Release (ER): 6-mg or 9-mg tablet once daily flexible dosing for 6 months
Period: Overall Study
Arm/Group | Paliperidone Extended Release (ER) | Olanzapine
Started | 239 | 220
Completed | 168 | 178
Not Completed | 71 | 42
Not completed — Lack of Efficacy | 15 | 6
Not completed — Withdrawal by Subject | 30 | 22
Not completed — Lost to Follow-up | 6 | 4
Not completed — Adverse Event | 11 | 5
Not completed — Other | 9 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paliperidone ER | Olanzapine | Total
Number analyzed (Participants) | 239 | 220 | 459
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (11.1) | 37.5 (11.4) | 38.2 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 87 | 193
  Male | 133 | 133 | 266
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 26.9 (6.31) | 27.0 (5.73) | 26.9 (6.03)
Waist [Mean (Standard Deviation); unit: cm] | 92.2 (14.4) | 93.3 (15.6) | 92.7 (14.9)
Weight [Mean (Standard Deviation); unit: kg] | 75.9 (17.0) | 77.9 (16.5) | 76.9 (16.8)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to End Point in the Triglycerides (TG) to High Density Lipoprotein (HDL) Ratio (TG:HDL Ratio)
Description: Plasma fasting TG and HDL concentrations were measured to determine the TG:HDL ratio.
Time Frame: Baseline to End Point (up to 6 months)
Population: The primary end point analysis set consisted of 413 patients, i.e., all patients who received study medication at least once and had baseline and post-baseline TG and HDL data. Data of patients with missing TG or HDL values or who started or changed lipid-lowering medication during the trial were excluded from analysis.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Paliperidone ER | Olanzapine
Number analyzed (Participants) | 215 | 198
Ratio | -0.08 (1.10) | 0.42 (1.19)
Statistical Analysis 1: Comparison: Paliperidone ER vs Olanzapine; Based on available data it was estimated that in the paliperidone ER group the TG:HDL ratio would decrease with 0.15 and that the TG:HDL ratio would increase with 0.25 in the olanzapine group. The common SD of the change was estimated to be 1.4. A sample size of 205 patients in each treatment arm had 80% power to detect a difference of 0.4 in change of TG:HDL ratio after 6 months of treatment in favor of paliperidone ER treatment (Wilcoxon two-sample test with 0.05 two-sided significance level); Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney); This test was interpreted at the 5% significance level (2-tailed)
Statistical Analysis 2: Comparison: Paliperidone ER; Within-group comparison of the change from baseline at end point; Test type: Superiority or Other; p = 0.4718, Wilcoxon signed rank test; This test was interpreted at the 5% significance level (2-tailed)
Statistical Analysis 3: Comparison: Olanzapine; Within-group change from baseline at end point; Test type: Superiority or Other; p < 0.0001, Wilcoxon signed rank test; This test was interpreted at the 5% significance level (2-tailed)

2. Secondary Outcome: Change From Baseline to End Point in Triglycerides
Description: The TG level was assessed under fasted conditions.
Time Frame: Baseline to End Point (up to 6 months)
Population: The secondary end point analysis set included all patients who received study medication at least once and provided ≥1 post-baseline efficacy measurement. Therefore, the total number of patients in the analysis set depends on the number of patients having post-baseline data for the particular secondary efficacy parameter under discussion.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Paliperidone ER | Olanzapine
Number analyzed (Participants) | 223 | 203
mmol/L | -0.01 (0.77) | 0.36 (0.96)
Statistical Analysis 1: Comparison: Paliperidone ER vs Olanzapine; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney); This test was interpreted at the 5% significance level (2-tailed)
Statistical Analysis 2: Comparison: Paliperidone ER; Within-group change from baseline to end point; Test type: Superiority or Other; p = 0.9143, Wilcoxon signed rank test; This test was interpreted at the 5% significance level (2-tailed)
Statistical Analysis 3: Comparison: Olanzapine; Within-group change from baseline to end point; Test type: Superiority or Other; p < 0.0001, Wilcoxon signed rank test; This test was interpreted at the 5% significance level (2-tailed)

3. Secondary Outcome: Change From Baseline to End Point in High Density Lipoprotein
Description: The HDL level was assessed under fasted conditions.
Time Frame: Baseline to End Point (up to 6 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Paliperidone ER | Olanzapine
Number analyzed (Participants) | 216 | 198
mmol/L | 0.01 (0.25) | -0.04 (0.24)
Statistical Analysis 1: Comparison: Paliperidone ER vs Olanzapine; Test type: Superiority or Other; p = 0.0050, Wilcoxon (Mann-Whitney); This test was interpreted at the 5% significance level (2-tailed)
Statistical Analysis 2: Comparison: Paliperidone ER; Within-group change from baseline to end point; Test type: Superiority or Other; p = 0.4454, Wilcoxon signed rank test; This test was interpreted at the 5% significance level (2-tailed)
Statistical Analysis 3: Comparison: Olanzapine; Within-group change from baseline to end point; Test type: Superiority or Other; p = 0.0018, Wilcoxon signed rank test; This test was interpreted at the 5% significance level (2-tailed)

4. Secondary Outcome: Change From Baseline to End Point in Total Cholesterol
Description: The total cholesterol level was assessed under fasted conditions.
Time Frame: Baseline to End Point (up to 6 months)
Population: Safety data were analyzed using the Intent-to-Treat (ITT) analysis set for safety and consisted of 459 patients, i.e., all patients who received study medication at least once and provided any post-baseline safety data. Changes from baseline could only be calculated for patients with paired data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Paliperidone ER | Olanzapine
Number analyzed (Participants) | 223 | 203
mmol/L | 0.0263 (0.7841) | 0.2886 (0.8493)
Statistical Analysis 1: Comparison: Paliperidone ER vs Olanzapine; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney); This test was interpreted at the 5% significance level (2-tailed)

5. Secondary Outcome: Change From Baseline to End Point in Low Density Lipoprotein Cholesterol (Friedwald QT)
Description: The level of low density lipoprotein cholesterol was calculated using the Friedwald QT formula.
Time Frame: Baseline to End Point (up to 6 months)
Population: Safety data were analyzed using the ITT analysis set for safety and consisted of 459 patients, i.e., all patients who received study medication at least once and provided any post-baseline safety data. Changes from baseline could only be calculated for patients with paired data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Paliperidone ER | Olanzapine
Number analyzed (Participants) | 216 | 194
mmol/L | -0.0029 (0.6726) | 0.1892 (0.7361)
Statistical Analysis 1: Comparison: Paliperidone ER vs Olanzapine; Test type: Superiority or Other; p = 0.0004, Wilcoxon (Mann-Whitney); This test was interpreted at the 5% significance level (2-tailed)

6. Secondary Outcome: Change From Baseline to End Point in Converted Insulin
Description: The insulin level was assessed under fasted conditions.
Time Frame: Baseline to End Point (up to 6 months)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Paliperidone ER | Olanzapine
Number analyzed (Participants) | 209 | 182
pmol/L | 2.7397 (89.9776) | 17.2327 (84.6255)
Statistical Analysis 1: Comparison: Paliperidone ER vs Olanzapine; Test type: Superiority or Other; p = 0.0272, Wilcoxon (Mann-Whitney); This test was interpreted at the 5% significance level (2-tailed)

7. Secondary Outcome: Change From Baseline to End Point in Fasting Glucose
Time Frame: Baseline to End Point (up to 6 months)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Paliperidone ER | Olanzapine
Number analyzed (Participants) | 14 | 13
mmol/L | -0.2071 (0.4953) | 0.0769 (0.4781)
Statistical Analysis 1: Comparison: Paliperidone ER vs Olanzapine; Test type: Superiority or Other; p = 0.1892, Wilcoxon (Mann-Whitney); This test was interpreted at the 5% significance level (2-tailed)

8. Secondary Outcome: Change From Baseline to End Point in Homeostatic Model Assessment of Beta-cell Function (HOMA-%B)
Description: HOMA-%B is used to assess beta-cell function. HOMA-%B is a dimensionless measure of beta-cell function (higher values present increased insulin secretion for a given glucose level).
  HOMA-%B is normalized so that lean, healthy individuals will have values of HOMA-%B close to 100%.
Time Frame: Baseline to End Point (up to 6 months)
Population: The secondary end point analysis set included all patients who received study medication at least once and provided ≥1 post-baseline efficacy measurement. Therefore, the total number of patients in the analysis set depends on the number of patients having post baseline data for the particular secondary efficacy parameter under discussion.
Measure: Mean (Standard Deviation); unit: dimensionless
Arm/Group | Paliperidone ER | Olanzapine
Number analyzed (Participants) | 183 | 174
dimensionless | -7.54 (85.91) | 18.82 (147.63)
Statistical Analysis 1: Comparison: Paliperidone ER vs Olanzapine; Test type: Superiority or Other; p = 0.0325, Wilcoxon (Mann-Whitney); This test was interpreted at the 5% significance level (2-tailed)

9. Secondary Outcome: Change From Baseline to End Point in Homeastatic Model Assessment of Insulin Resistance (HOMA-IR)
Description: HOMA-IR is used to assess insulin resistance (IR). HOMA-IR is a dimensionless measure of insulin resistance (higher values present more insulin resistance. HOMA-IR are normalized so that lean, healthy individuals will have values of HOMA-IR close to 1.
Time Frame: Baseline to End Point (up to 6 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: dimensionless
Arm/Group | Paliperidone ER | Olanzapine
Number analyzed (Participants) | 184 | 174
dimensionless | 0.28 (5.39) | 0.43 (5.37)
Statistical Analysis 1: Comparison: Paliperidone ER vs Olanzapine; Test type: Superiority or Other; p = 0.1117, Wilcoxon (Mann-Whitney); This test was interpreted at the 5% significance level (2-tailed)

10. Secondary Outcome: Number of Patients Meeting the Criteria for Type 2 Diabetes Mellitus During Follow-up
Description: Fasting plasma glucose ≥126 mg/dL or 2-hour post-load plasma glucose ≥200 mg/dL during an oral glucose tolerance test (OGTT) or initiated use of glucose-lowering agents during the course of the study.
Time Frame: 6 months
Population: The secondary end point analysis set included all patients who received study medication at least once and provided ≥1 post-baseline efficacy measurement.Therefore, the total number of patients in the analysis set depends on the number of patients having post-baseline data for the particular secondary efficacy parameter under discussion.
Measure: Number; unit: Participants
Arm/Group | Paliperidone ER | Olanzapine
Number analyzed (Participants) | 239 | 220
Participants | 21 | 23
Statistical Analysis 1: Comparison: Paliperidone ER vs Olanzapine; Test type: Superiority or Other; p = 0.6346, Fisher Exact; This test was interpreted at the 5% significance level (2-tailed)

11. Secondary Outcome: Number of Patients With Onset of Impaired Glucose Tolerance
Description: Glucose ≥140 mg/dL, <200 mg/dL after a 75g OGTT.
Time Frame: Baseline to End Point (up to 6 months)
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | Paliperidone ER | Olanzapine
Number analyzed (Participants) | 217 | 198
Participants | 36 | 33
Statistical Analysis 1: Comparison: Paliperidone ER vs Olanzapine; Test type: Superiority or Other; p = 1.0000, Fisher Exact; This test was interpreted at the 5% significance level (2-tailed)

12. Secondary Outcome: Number of Patients With Impaired Fasting Glucose
Description: Post-baseline glucose level under fasted conditions ≥100 mg/dL but <126 mg/dL.
Time Frame: Baseline to End Point (up to 6 months)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Paliperidone ER | Olanzapine
Number analyzed (Participants) | 223 | 203
Participants | 68 | 66
Statistical Analysis 1: Comparison: Paliperidone ER vs Olanzapine; Test type: Superiority or Other; p = 0.6770, Fisher Exact; This test was interpreted at the 5% significance level (2-tailed)

13. Secondary Outcome: Change From Baseline at End Point of the Insulinogenic Index
Description: The insulinogenic index, defined as (insulin at 30 min - insulin at 0)/(glucose at 30 min [G(30)] - glucose at 0 [G(0)]) was used as a measure of early insulin secretion in response to the OGTT. Because the index is undefined when G(30)-G(0)=0, and poorly defined when G(30)-G(0)<0, the index was only calculated when G(30)>G(0).
Time Frame: Baseline to End Point (up to 6 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pM/mM
Arm/Group | Paliperidone ER | Olanzapine
Number analyzed (Participants) | 154 | 147
pM/mM | 2.21 (173.46) | 33.78 (259.56)
Statistical Analysis 1: Comparison: Paliperidone ER vs Olanzapine; Test type: Superiority or Other; p = 0.1308, Wilcoxon (Mann-Whitney); This test was interpreted at the 5% significance level (2-tailed)

14. Secondary Outcome: Change From Baseline at End Point of Mari-Type Analysis of Glucose Sensitivity for Insulin
Description: As another measure of beta-cell function, the relationship between plasma insulin and glucose concentrations during the OGTT was calculated using a simplified version of the method described by Mari et al. (Mari A, Sallas WM, He YL, Watson C, Ligueros-Saylan M, Dunning BE, Deacon CF, Holst JJ, Foley JE. Vildagliptin, a dipeptidyl peptidase-IV inhibitor, improves model-assessed beta-cell function in patients with type 2 diabetes. J Clin Endocrinol Metab. 2005; 90:4888-4894.).
Time Frame: Baseline to End Point (up to 6 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pM/mM
Arm/Group | Paliperidone ER | Olanzapine
Number analyzed (Participants) | 183 | 169
pM/mM | 8.63 (79.53) | 17.28 (94.51)
Statistical Analysis 1: Comparison: Paliperidone ER vs Olanzapine; Test type: Superiority or Other; p = 0.3358, Wilcoxon (Mann-Whitney); This test was interpreted at the 5% significance level (2-tailed)

15. Secondary Outcome: Change From Baseline at End Point in Body Weight
Description: Patients were weighed lightly clothed. The same amount of clothing had to be worn each time.
Time Frame: Baseline to End Point (up to 6 months)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Paliperidone ER | Olanzapine
Number analyzed (Participants) | 235 | 214
kg | 1.16 (4.57) | 3.81 (5.87)
Statistical Analysis 1: Comparison: Paliperidone ER vs Olanzapine; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney); This test was interpreted at the 5% significance level (2-tailed)
Statistical Analysis 2: Comparison: Paliperidone ER; Within-group change from baseline to end point; Test type: Superiority or Other; p = 0.0001, Wilcoxon signed rank test; This test was interpreted at the 5% significance level (2-tailed)
Statistical Analysis 3: Comparison: Olanzapine; Within-group change from baseline to end point; Test type: Superiority or Other; p < 0.0001, Wilcoxon signed rank test; This test was interpreted at the 5% significance level (2-tailed)

16. Secondary Outcome: Change From Baseline at End Point in Body Mass Index (BMI)
Description: BMI is calculated by dividing the body weight (in kg) by the square of height (in meters).
Time Frame: Baseline to End Point (up to 6 months)
Measure: Mean (Standard Deviation); unit: kg/m²
Arm/Group | Paliperidone ER | Olanzapine
Number analyzed (Participants) | 235 | 214
kg/m² | 0.43 (1.59) | 1.32 (1.99)
Statistical Analysis 1: Comparison: Paliperidone ER vs Olanzapine; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney); This test was interpreted at the 5% significance level (2-tailed)

17. Secondary Outcome: Change From Baseline at End Point in Waist Circumference
Description: Patients had to be instructed to stand erect with abdomen relaxed, arms at sides, feet together, and weight divided equally over both legs. The tape measure was placed around the bare abdomen midway between the palpated iliac crest and the palpated lowest rib margin in the left and right mid-axillary lines. A nonstretchable tape was evenly placed around the natural waist covering the left and right natural-waist marks. The measurement scale had to face outward, and there could not be any twists in the tape. The tape had to be just touching the skin but not compressing the soft tissue.
Time Frame: Baseline to End Point (up to 6 months)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Paliperidone ER | Olanzapine
Number analyzed (Participants) | 231 | 213
cm | 0.70 (5.39) | 3.38 (6.18)
Statistical Analysis 1: Comparison: Paliperidone ER vs Olanzapine; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney); This test was interpreted at the 5% significance level (2-tailed)

18. Secondary Outcome: Number of Patients First Meeting the NCEP/ATP III Criteria for Metabolic Syndrome During Follow-up
Description: Metabolic syndrome is defined according the Third Report of the National Cholesterol Education Program Expert Panel on
  Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (NCEP/ATPIII) of which 3 out of 5 criteria must be met:
  * waist circumference men > 102 cm; waist circumference women > 88 cm
  * TG ≥ 150 mg/dL
  * HDL cholesterol men <40 mg/dL; HDL cholesterol women <50 mg/dL
  * Blood pressure systolic ≥ 130 mmHg; Blood pressure diastolic ≥ 85 mmHg
  * Fasting glucose ≥ 110 mg /dL
Time Frame: 6 months
Population: The secondary endpoint analysis set included all patients who received study medication at least once and provided ≥1 post-baseline efficacy measurement. In this case, the total number of patients in the analysis set depends on the number of patients without metabolic syndrome at baseline.
Measure: Number; unit: Participants
Arm/Group | Paliperidone ER | Olanzapine
Number analyzed (Participants) | 174 | 163
Participants | 23 | 38
Statistical Analysis 1: Comparison: Paliperidone ER vs Olanzapine; Test type: Superiority or Other; p = 0.0230, Fisher Exact; This test was interpreted at the 5% significance level (2-tailed)

19. Secondary Outcome: Change From Baseline to End Point in Total Positive and Negative Syndrome Scale Score (PANSS)
Description: PANSS is an investigator-rated 30-item scale to assess the neuropsychiatric symptoms of schizophrenia. The PANSS provided a total score and scores for 3 subscales, the positive subscale (7 items), the negative subscale (7 items), and the general psychopathology subscale (16 items), each rated on a scale of 1 (absent) to 7 (extreme).
Time Frame: Baseline to End Point (up to 6 months)
Population: The secondary endpoint analysis set included all patients who received study medication at least once and provided ≥1 post-baseline efficacy measurement. Therefore, the total number of patients in the analysis set depends on the number of patients having post-baseline data for the particular secondary efficacy parameter under discussion.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Paliperidone ER | Olanzapine
Number analyzed (Participants) | 234 | 214
points on a scale | -13.50 (15.86) | -16.60 (15.02)
Statistical Analysis 1: Comparison: Paliperidone ER vs Olanzapine; Test type: Non-Inferiority or Equivalence — Testing non-inferiority of the paliperidone ER treatment group compared to the olanzapine treatment group, with regard to change versus baseline at end point of the total PANSS was done by means of Schuirmann's test. A difference of 6 points in change versus baseline on the total PANSS was considered to be a minimum clinically relevant difference.The null hypothesis is that there is no difference between paliperidone and olanzapine in change in TG:HDL ratio from baseline to endpoint; p = 0.0242, Schuirmann; The null hypothesis of non-equivalence was rejected and equivalence to within the specified equivalence bounds could be claimed
Statistical Analysis 2: Comparison: Paliperidone ER; Within-group change from baseline to end point; Test type: Superiority or Other; p < 0.0001, Wilcoxon signed rank test; This test was interpreted at the 5% significance level (2-tailed)
Statistical Analysis 3: Comparison: Olanzapine; Within-group change from baseline to end point; Test type: Superiority or Other; p < 0.0001, Wilcoxon signed rank test; This test was interpreted at the 5% significance level (2-tailed)

ADVERSE EVENTS:
Time Frame: From informed consent up to 6 months (+/- 7 days) of treatment. In case subjects had discontinued before completing treatment, the last data were obtained at the early discontinuation visit.
Arm/Group | Paliperidone ER | Olanzapine
Serious Adverse Events (participants affected / at risk) | 21/239 | 12/220
Other Adverse Events (participants affected / at risk) | 98/239 | 93/220
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone ER (N=239) | Olanzapine (N=220)
Schizophrenia (Psychiatric disorders) | 8 | 3
Psychotic disorder (Psychiatric disorders) | 6 | 1
Depression (Psychiatric disorders) | 2 | 0
Psychiatric decompensation (Psychiatric disorders) | 0 | 2
Psychiatric symptom (Psychiatric disorders) | 1 | 1
Intentional self-injury (Psychiatric disorders) | 1 | 0
Nervousness (Psychiatric disorders) | 0 | 1
Schizophrenia, paranoid type (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Mastitis (Infections and infestations) | 0 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone ER (N=239) | Olanzapine (N=220)
Weight increased (Investigations) | 23 | 40
Blood creatine phosphokinase increased (Investigations) | 7 | 5
Alanine aminotransferase increased (Investigations) | 1 | 3
Blood glucose increased (Investigations) | 1 | 3
Gamma-glutamyltransferase increased (Investigations) | 1 | 3
Waist circumference increased (Investigations) | 0 | 4
Weight decreased (Investigations) | 3 | 1
Blood triglycerides increased (Investigations) | 0 | 3
Somnolence (Nervous system disorders) | 8 | 21
Headache (Nervous system disorders) | 11 | 9
Sedation (Nervous system disorders) | 5 | 6
Akathisia (Nervous system disorders) | 6 | 2
Dizziness (Nervous system disorders) | 5 | 2
Dyskinesia (Nervous system disorders) | 3 | 2
Hypersomnia (Nervous system disorders) | 3 | 2
Insomnia (Psychiatric disorders) | 23 | 3
Anxiety (Psychiatric disorders) | 10 | 3
Tension (Psychiatric disorders) | 5 | 1
Agitation (Psychiatric disorders) | 4 | 1
Schizophrenia (Psychiatric disorders) | 4 | 1
Psychotic disorder (Psychiatric disorders) | 3 | 1
Restlessness (Psychiatric disorders) | 3 | 1
Depression (Psychiatric disorders) | 0 | 3
Fatigue (General disorders) | 5 | 2
Irritability (General disorders) | 3 | 3
Influenza (Infections and infestations) | 2 | 3
Nasopharyngitis (Infections and infestations) | 3 | 1
Urinary tract infection (Infections and infestations) | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 4 | 2
Nausea (Gastrointestinal disorders) | 3 | 1
Amenorrhoea (Reproductive system and breast disorders) | 8 | 0
Galactorrhoea (Reproductive system and breast disorders) | 3 | 0
Increased appetite (Metabolism and nutrition disorders) | 4 | 5
Hypertension (Vascular disorders) | 2 | 3
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3 | 0

LIMITATIONS AND CAVEATS:
Open-label design

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days